CLINICAL TRIAL: NCT04443959
Title: Telemedicine Mindfulness-based Therapy for Perinatal Insomnia: An Open-label Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, David Kalmbach, Bioscientific Staff Researcher, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPD2
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Insomnia
Keywords: Mindfulness; Cognitive arousal; insomnia; pregnant; perinatal
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PUMAS Treatment (Experimental): Prenatal insomnia program that places behavioral sleep strategies within a mindfulness-based intervention framework that is geared toward pregnant women.
  Interventions: Behavioral: PUMAS

INTERVENTIONS:
Behavioral: PUMAS — Treatment consists of 6 weekly telemedicine sessions during pregnancy.

SUMMARY:
Over half of pregnant and postpartum women experience clinical insomnia. However, treatment options are very limited for pregnant women and moms of newborns. Sleep aids are not considered safe during pregnancy and may increase risks about safety for mom and baby during postpartum. Recent clinical trials show that behavioral and mindfulness-based treatments can safely improve sleep and mood during pregnancy. Yet, no published studies to date have combined behavioral sleep treatment with mindfulness-based stress reduction to improve sleep and mood at the same time in pregnant and postpartum women. This study is the first to combine behavioral sleep strategies with mindfulness-meditation to improve sleep and psychological wellbeing of expecting and new moms.

The purpose of this research study is to examine the effectiveness of a mindfulness-based intervention for prenatal insomnia via telemedicine format to improve sleep and mood as well as reduce stress in pregnant women.

DETAILED DESCRIPTION:
The purpose of this open-label trial is to determine the efficacy of and patient engagement in mindfulness-based intervention for prenatal insomnia delivered via telemedicine. The investigators' long-term goal is to improve sleep and mood of expecting and new mothers. Over half of pregnant women develop insomnia, which is associated with high rates of depression during pregnancy and postpartum. By successfully treating insomnia during pregnancy and improving cognitive-emotion regulation, mental health of pregnant women and new moms may be greatly improved. In a prior clinical trial, Dr. Kalmbach (PI) showed that online cognitive-behavioral therapy for insomnia (CBTI) greatly improved sleep during pregnancy, and offered some protection against sleep problems after childbirth. Women in this trial were highly satisfied with CBTI and especially its remote delivery. However, the investigators identified important shortcomings of online CBTI in this population. Namely, patients provided feedback that reducing cognitive arousal (ie ruminative or worrisome thinking) was an important therapeutic target, that more mindfulness-based approaches and strategies would improve treatment, and that greater emphasis on maternal and infant sleep would also enhance the treatment experience. Thus, the investigators will conduct an open label trial to collect pilot data on the efficacy of a telemedicine mindfulness-based intervention for prenatal insomnia that has been tailored for pregnant women. Specifically, the investigators will conduct this open-label trial of 50 pregnant women to preliminary test the efficacy, patient adherence, patient engagement, and patient satisfaction with this telemedicine program.

This open-label trial will enroll 50 pregnant women (gestational age 18-30 weeks at study entry) who will receive 6 sessions of 'Perinatal Understanding of Mindful Awareness for Sleep' (PUMAS) via telemedicine video with a therapist. Patients will complete this treatment during pregnancy. This program was based on Dr. Jason Ong's Mindfulness-Based Therapy for Insomnia, which combined CBTI and mindfulness meditation, and it has been tailored for perinatal women. The investigators will assess study outcomes before treatment and after treatment. Study outcomes will include insomnia symptoms, depressive symptoms, and cognitive arousal. The investigators will also assess patient engagement (number of completed sessions, homework adherence) and collect patient feedback (e.g., treatment satisfaction).

ELIGIBILITY:
Inclusion Criteria:

* (1) Gestational age at time of study enrollment must be 18-30 weeks.
* (2) Insomnia Severity Index score of 11 or higher
* (3) age between 18 and 40 years
* (4) reliable and adequately fast internet connection at home, which is required to engage in online treatment and online study outcome assessments

Exclusion Criteria:

* (1) High risk pregnancy as reported by the patient, which includes but is not limited to pre-eclampsia, gestational diabetes, maternal age > 40, ectopic pregnancy, fetal problems (e.g., heart problems), hyperemesis gravidarum, placenta previa, and placental abruption.
* (2) bipolar disorder or seizure disorders [contraindicated for insomnia therapy] as reported by the patient
* (3) women with multiple pregnancy (e.g., twins, triplets, etc.) will not be eligible to participate as multiple pregnancy can increase risk of complications and often leads to preterm or early-term birth
* (4) any conditions or difficulties that would prevent the patient from completing online treatment and/or online surveys, including but not limited to language difficulties, literacy issues, visual or auditory impairment, and cognitive deficits
* (5) active suicidal intent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Effectiveness of PUMAS for changes in insomnia symptoms - Insomnia Severity Index (ISI) | Pretreatment, then posttreatment (after completing prenatal treatment or 10 weeks after starting prenatal treatment).
  The Insomnia Severity Index (ISI) is a commonly used self-report measure of insomnia symptoms that has been validated for use in community samples and clinical trials. The ISI scores range from 0-28, with a higher score indicating a greater severity of insomnia. ISI scores < 8 after treatment indicate remission.

SECONDARY OUTCOMES:
Effectiveness of PUMAS for changes in depressive symptoms | Pretreatment, then posttreatment (after completing prenatal treatment or 10 weeks after starting prenatal treatment).
  The Edinburgh Postnatal Depression (EPDS) is the most widely used depression measure in both pregnant and postnatal women. It is validated for use in community samples and clinical trials. The EPDS scores range from 0-30, with a higher score indicating a greater severity of depression.
Effectiveness of PUMAS for changes in of cognitive arousal- Presleep Arousal Scale- Cognitive Factor | Pretreatment, then posttreatment (after completing prenatal treatment or 10 weeks after starting prenatal treatment).
  The Presleep Arousal Scale - Cognitive Factor is a commonly used self-report measure of insomnia symptoms that has been validated for use in community samples and clinical trials. The scores range from 8-40, with a higher score indicating a greater severity of nocturnal cognitive arousal.

CONTACTS AND LOCATIONS:
Overall Officials: David Kalmbach, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Medical Center, Novi, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kalmbach DA, Cheng P, Reffi AN, Ong JC, Swanson LM, Espie CA, Seymour GM, Hirata M, Walch O, Pitts DS, Roth T, Drake CL. Reducing cognitive arousal and sleep effort alleviates insomnia and depression in pregnant women with DSM-5 insomnia disorder treated with a mindfulness sleep program. Sleep Adv. 2023 Aug 5;4(1):zpad031. doi: 10.1093/sleepadvances/zpad031. eCollection 2023. PMID 37645455
- [Derived] Kalmbach DA, Cheng P, Reffi AN, Ong JC, Swanson LM, Fresco DM, Walch O, Seymour GM, Fellman-Couture C, Bayoneto AD, Roth T, Drake CL. Perinatal Understanding of Mindful Awareness for Sleep (PUMAS): A single-arm proof-of-concept clinical trial of a mindfulness-based intervention for DSM-5 insomnia disorder during pregnancy. Sleep Med. 2023 Aug;108:79-89. doi: 10.1016/j.sleep.2023.05.026. Epub 2023 Jun 10. PMID 37343335